CLINICAL TRIAL: NCT06839794
Title: An Investigator Initiated, Non-randomized Controlled Trial on the Effect of Cognitively Challenging Physical Activity on Executive Functions in Paediatric Cancer Patients
Brief Title: Effect of Cognitively Challenging Physical Activity on Executive Functions in Pediatric Cancer Patients
Acronym: KiKli Fit
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other); University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-00923
Record Dates: First submitted 2025-02-10; First posted 2025-02-21 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Childhood Cancer; Cancer-related Problem/Condition; Cognitive Side Effects of Cancer Therapy; Physical Activity
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: During the first phase, the intervention will commence at the Inselspital Bern, and the University Children's Hospital Basel and Aarau will serve as the control. In the second phase, after 1.5 years, a crossover will take place, and Bern will serve as the control, while the intervention takes place in Basel and Aarau.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Intervention (Other): Participants have access to standard care as usual and receive physical activity recommendations.
  Interventions: Other: Physical activity recommendations
- Intervention (Experimental): The intervention is a cognitively challenging physical activity (PA) intervention for children and adolescents with cancer undergoing acute therapy. The intervention is based on the "S2k Guideline: Promotion of Exercise and Exercise Therapy in Paediatric Oncology" and the international Paediatric Oncology Exercise Guidelines. And on study results and experience from previous cognitive challenging PA intervention studies.
  Interventions: Behavioral: Cognitively challenging physical activity for paediatric cancer patients

INTERVENTIONS:
Behavioral: Cognitively challenging physical activity for paediatric cancer patients — The intervention is a structured cognitively challenging physical activity (PA) program specifically designed for pediatric cancer patients undergoing acute therapy. It stands out from other interventions by combining motor and cognitive tasks simultaneously. Therefore, the target executive functions are inhibition, shifting, and updating. Additionally, the whole body is addressed by enhancing PA.
  The PA program spans 12 weeks, with each participant engaging in guided, supervised 45-minute sessions three times weekly. Each session includes a warm-up, the cognitive challenging PA task and a subsequent multimodal sports programme with a cool-down. Exercises are adaptive and tailored to each participant's physical and health condition by offering three levels of intensity in both cognitive and physical difficulty. In addition, exercise counselling in maintenance therapy or aftercare supports young patients to reintegrate into the life after the disease.
  Other Names: KiKli Fit Study
  Arms: Intervention
Other: Physical activity recommendations — The children and adolescents receive general physical activity recommendations at the baseline measurement (t0). At the end of the intervention (after 12 weeks), i.e. after the final measurement (t3), they receive individualised and tailored exercise recommendations based on the test results from t0-t3.
  Arms: Control Intervention

SUMMARY:
When it comes to exercise and sport for children and adolescents with cancer, there is often still the opinion that physical activity has a negative effect on the weakened body suffering from cancer. Many studies show that the opposite is the case: physical activity for children and adolescents with cancer do not jeopardise the success of treatment, but rather promote it. It has been shown that physical activity has a positive effect on motor skills, physical fitness, sleep quality, fatigue symptoms, body image and general quality of life in children and adolescents with cancer.

In addition, physical activity leads to an improved fat-to-muscle ratio, metabolic status, bone strength and reduces cardiovascular disease. Furthermore, various studies show that oncological patients with sarcopenia (loss of muscle mass) and frailty have a poorer response to their cancer therapy. This broad spectrum of effects of physical activity leads to improved and faster rehabilitation, is directly linked to the success of treatment and has led to exercise being an integral part of treatment in many paediatric oncology centres worldwide.

Furthermore, more exercise that includes playful cognitive tasks is expected to lead to improved attention, memory and academic achievement. Besides, it is important to try to get children to exercise at home outside of the inpatient setting. Hybrid (on-site and digital meetings) programmes also work for children and adolescents. Additionally, the research project offers sports counselling after the end of therapy to reintegrate the patients into everyday sporting life, be it in a club or at school.

The central question of the research project is: Does cognitive challenging physical activity developed for children and adolescents undergoing acute cancer therapy improve cognitive and motor performance compared to a control group receiving standard care?

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of parents / legal guardian and participants, where applicable
* Diagnosis of any type of cancer requiring chemo- and/or radiotherapy, or CNS surgery, expected to last a minimum of at least 6 weeks at the time of recruitment
* Age: 6-17.99 years at time of recruitment

Exclusion Criteria:

* Cognitive and physical disabilities that prevent participation in the intervention.
* Inability to follow the procedures of the study, e.g. due to language problems.
* Enrolment of the investigator, his/her family members, employees and other dependent persons.
* Denied written informed consent from participants.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2025-05-10 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Executive function, assessed via Hearts and Flowers Task | Baseline measurement around the first 3 weeks after diagnosis
  The Hearts and Flowers Task is a cognitive test designed to measure executive functions, particularly inhibitory control and cognitive flexibility. The test consists of two types of conditions: In the simple condition (hearts), participants are instructed to respond on the same side as the heart appears. In the complex condition (flowers), they are instructed to respond on the opposite side of the flower's appearance. Reaction time and accuracy are recorded.
Executive function, assessed via Hearts and Flowers Task | Interim measurement (T1) 6 weeks after baseline
  The Hearts and Flowers Task is a cognitive test designed to measure executive functions, particularly inhibitory control and cognitive flexibility. The test consists of two types of conditions: In the simple condition (hearts), participants are instructed to respond on the same side as the heart appears. In the complex condition (flowers), they are instructed to respond on the opposite side of the flower's appearance. Reaction time and accuracy are recorded.
Executive function, assessed via Hearts and Flowers Task | Post assessment measurement (T2) 12 weeks after baseline
  The Hearts and Flowers Task is a cognitive test designed to measure executive functions, particularly inhibitory control and cognitive flexibility. The test consists of two types of conditions: In the simple condition (hearts), participants are instructed to respond on the same side as the heart appears. In the complex condition (flowers), they are instructed to respond on the opposite side of the flower's appearance. Reaction time and accuracy are recorded.
Executive function, assessed via Hearts and Flowers Task | Follow-up measurement (T3) 6 month after baseline
  The Hearts and Flowers Task is a cognitive test designed to measure executive functions, particularly inhibitory control and cognitive flexibility. The test consists of two types of conditions: In the simple condition (hearts), participants are instructed to respond on the same side as the heart appears. In the complex condition (flowers), they are instructed to respond on the opposite side of the flower's appearance. Reaction time and accuracy are recorded.
Executive function, assessed via Fish-Flanker Task | Baseline measurement around the first 3 weeks after diagnosis
  The Fish-Flanker Task is a cognitive test used to measure inhibitory control. Participants are shown a row of five fish and must respond to the direction of the central target fish while ignoring the surrounding flanker fish. In congruent trials, the flankers face the same direction as the target fish, while in incongruent trials, they face the opposite direction. Reaction time and accuracy are recorded.
Executive function, assessed via Fish-Flanker Task | Interim measurement (T1) 6 weeks after baseline
  The Fish-Flanker Task is a cognitive test used to measure inhibitory control. Participants are shown a row of five fish and must respond to the direction of the central target fish while ignoring the surrounding flanker fish. In congruent trials, the flankers face the same direction as the target fish, while in incongruent trials, they face the opposite direction. Reaction time and accuracy are recorded.
Executive function, assessed via Fish-Flanker Task | Post assessment measurement (T2) 12 weeks after baseline
  The Fish-Flanker Task is a cognitive test used to measure inhibitory control. Participants are shown a row of five fish and must respond to the direction of the central target fish while ignoring the surrounding flanker fish. In congruent trials, the flankers face the same direction as the target fish, while in incongruent trials, they face the opposite direction. Reaction time and accuracy are recorded.
Executive function, assessed via Fish-Flanker Task | Follow-up measurement (T3) 6 month after baseline
  The Fish-Flanker Task is a cognitive test used to measure inhibitory control. Participants are shown a row of five fish and must respond to the direction of the central target fish while ignoring the surrounding flanker fish. In congruent trials, the flankers face the same direction as the target fish, while in incongruent trials, they face the opposite direction. Reaction time and accuracy are recorded.
Executive function, assessed via Corsi Block Task | Baseline measurement around the first 3 weeks after diagnosis
  The Corsi Block Task is a cognitive test used to measure visuospatial working memory. Participants are shown a series of blocks on a screen, which light up in a specific sequence. The task requires replicating the sequence by tapping the blocks in the same order (forward condition) or in reverse order (backward condition). The length of the sequence increases after each correct attempt. The score is the longest correctly repeated sequence, ranging from 0 (no correct sequences) to 10 or more (longer sequences).
  The outcome measures include the total number of correctly recalled sequences, the achieved Block Span, the z-score of the Block Span and the percentile of the Block Span. Additionally, they include a summary score calculated as the product of the Block Span and the total number of correct sequences, the z-score of this total score and the percentile of the total score.
Executive function, assessed via Corsi Block Task | Interim measurement (T1) 6 weeks after baseline
  The Corsi Block Task is a cognitive test used to measure visuospatial working memory. Participants are shown a series of blocks on a screen, which light up in a specific sequence. The task requires replicating the sequence by tapping the blocks in the same order (forward condition) or in reverse order (backward condition). The length of the sequence increases after each correct attempt. The score is the longest correctly repeated sequence, ranging from 0 (no correct sequences) to 10 or more (longer sequences).
  The outcome measures include the total number of correctly recalled sequences, the achieved Block Span, the z-score of the Block Span and the percentile of the Block Span. Additionally, they include a summary score calculated as the product of the Block Span and the total number of correct sequences, the z-score of this total score and the percentile of the total score.
Executive function, assessed via Corsi Block Task | Post assessment measurement (T2) 12 weeks after baseline
  The Corsi Block Task is a cognitive test used to measure visuospatial working memory. Participants are shown a series of blocks on a screen, which light up in a specific sequence. The task requires replicating the sequence by tapping the blocks in the same order (forward condition) or in reverse order (backward condition). The length of the sequence increases after each correct attempt. The score is the longest correctly repeated sequence, ranging from 0 (no correct sequences) to 10 or more (longer sequences).
  The outcome measures include the total number of correctly recalled sequences, the achieved Block Span, the z-score of the Block Span and the percentile of the Block Span. Additionally, they include a summary score calculated as the product of the Block Span and the total number of correct sequences, the z-score of this total score and the percentile of the total score.
Executive function, assessed via Corsi Block Task | Follow-up measurement (T3) 6 month after baseline
  The Corsi Block Task is a cognitive test used to measure visuospatial working memory. Participants are shown a series of blocks on a screen, which light up in a specific sequence. The task requires replicating the sequence by tapping the blocks in the same order (forward condition) or in reverse order (backward condition). The length of the sequence increases after each correct attempt. The score is the longest correctly repeated sequence, ranging from 0 (no correct sequences) to 10 or more (longer sequences).
  The outcome measures include the total number of correctly recalled sequences, the achieved Block Span, the z-score of the Block Span and the percentile of the Block Span. Additionally, they include a summary score calculated as the product of the Block Span and the total number of correct sequences, the z-score of this total score and the percentile of the total score.

SECONDARY OUTCOMES:
Self-regulation, assessed via Head-Toes-Knees-Shoulders-task | Baseline measurement around the first 3 weeks after diagnosis; interim measurement (T1) 6 weeks after baseline; post assessment measurement (T2) 12 weeks after baseline; follow-up measurement (T3) 6 month after baseline
  Self-regulation will be assessed using the Head-Toes-Knees-Shoulders task (HTKS). This task measures self-regulation by requiring participants to follow specific instructions that conflict with automatic responses.
  The task involves a series of instructions where participants are asked to perform actions that oppose their natural impulses. For example, they may be asked to touch their head when instructed to touch their toes or to touch their knees when told to touch their shoulders.
  For a wrong movement the participant gets 0, for a corrected movement 1 and for a correct movement 2 points.
  The score ranges from 0-60.
Frailty, assessed via Frailty Score | Baseline measurement around the first 3 weeks after diagnosis; interim measurement (T1) 6 weeks after baseline; post assessment measurement (T2) 12 weeks after baseline; follow-up measurement (T3) 6 month after baseline
  The frailty score is calculated to assess an individual's vulnerability and considering 5 different aspects.
  Weakness, slowness, shrinkage, exhaustion and diminished physical activity. These are defined by the following corresponding parameters, the hand strength measurement from the Moon Test, the 6 MWT, the triceps skinfold thickness, the PedsQL fatigue scale, as well as the PedsQL core and the BSA as well as the Godin-Shephard Leisure-Time Physical Activity Questionnaire (GSLTPAQ). All tests are already listed and described in the outcomes.
  The frailty score is the composite endpoint of the named tests. The score ranges from 0 to 10, with a higher value indicating greater frailty (meaning higher Frailty worse clinical outcome).
Cardiovascular Health, assessed via Heart Rate Variability (HRV) | Baseline measurement around the first 3 weeks after diagnosis; interim measurement (T1) 6 weeks after baseline; post assessment measurement (T2) 12 weeks after baseline; follow-up measurement (T3) 6 month after baseline
  Heart rate variability (HRV) will be assessed using an ECG 4 activity sensor. HRV provides insights into how the heart responds to stress and relaxation. A high HRV is typically associated with better cardiovascular fitness, a more adaptable autonomic nervous system, and greater resilience to stress. Conversely, low HRV is often linked to poor health outcomes, such as higher stress levels, cardiovascular issues, and an increased risk of chronic diseases. Monitoring HRV can help assess an individual's overall well-being and autonomic nervous system functioning, as well as their response to various stressors.
Cardiovascular Health, assessed via Aortic Stiffness | Baseline measurement around the first 3 weeks after diagnosis; interim measurement (T1) 6 weeks after baseline; post assessment measurement (T2) 12 weeks after baseline; follow-up measurement (T3) 6 month after baseline
  Aortic Stiffness will be measured with the Mobil-O-Graph. This test helps to understand how flexible or stiff the aorta is, which is important for blood flow and blood pressure. Aortic stiffness is a key indicator of cardiovascular health, as it reflects the ability of the aorta to expand and contract with each heartbeat. Increased stiffness of the aorta can lead to higher systolic blood pressure and can be a risk factor for cardiovascular diseases.
Cardiovascular Health, assessed via 6-Minute Walk Test | Baseline measurement around the first 3 weeks after diagnosis; interim measurement (T1) 6 weeks after baseline; post assessment measurement (T2) 12 weeks after baseline; follow-up measurement (T3) 6 month after baseline
  The cardiopulmonary function will be evaluated with the 6-Minute Walk Test (6MWT). This test measures overall endurance and heart-lung efficiency by walking as fast as possible for 6 minutes. A longer distance walked in 6 minutes generally indicates better cardiovascular and pulmonary health, while shorter distances may signal reduced endurance or impaired heart-lung function. The test is particularly useful for evaluating patients with cardiovascular and respiratory conditions, as it provides an objective measure of physical capability and helps track changes in health status over time.
Body composition, assessed via Triceps Skin-Fold Thickness | Baseline measurement around the first 3 weeks after diagnosis; interim measurement (T1) 6 weeks after baseline; post assessment measurement (T2) 12 weeks after baseline; follow-up measurement (T3) 6 month after baseline
  Triceps skin-fold thickness will be measured with calipers to estimate body fat percentage based on the thickness of the skinfold at the triceps. This will be needed to calculate the frailty score.
Health-Related Quality of Life, assessed via PedsQL | Baseline measurement around the first 3 weeks after diagnosis; interim measurement (T1) 6 weeks after baseline; post assessment measurement (T2) 12 weeks after baseline; follow-up measurement (T3) 6 month after baseline
  Health-related Quality of Life (HrQoL) will be assessed with the Pediatric Quality of Life Inventory (PedsQL 4.0 Generic Core Scales), which measures overall well-being and quality of life.
  The score ranges from 0-100. Higher scores signifying better HrQoL.
Cancer related fatigue, assessed via PedsQL Fatigue Module | Baseline measurement around the first 3 weeks after diagnosis; interim measurement (T1) 6 weeks after baseline; post assessment measurement (T2) 12 weeks after baseline; follow-up measurement (T3) 6 month after baseline
  Cancer-related fatigue will be assessed with the PedsQL Fatigue Module. This questionnaire is designed to evaluate fatigue in pediatric populations, including its impact on physical, emotional, and cognitive functioning. Scores are reversed and linearly transformed to a scale of 0 to 100, where higher scores indicate less fatigue and better functioning. Subscale scores and a total fatigue score can be calculated by averaging the item responses, providing a comprehensive assessment of fatigue levels.
Physical Self-Concept, assessed via PSDQ-S | Baseline measurement around the first 3 weeks after diagnosis; interim measurement (T1) 6 weeks after baseline; post assessment measurement (T2) 12 weeks after baseline; follow-up measurement (T3) 6 month after baseline
  Physical Self-Concept will be measured with the Physical Self-Description Questionnaire - short version (PSDQ-S), focusing on how participants view their physical abilities.
  The questionnaire contains 22 questions. The score reaches from 22-132. The higher the score the greater the clinical outcome and physical self-concept.
Physical Activity Enjoyment, assessed via PACES-S | Baseline measurement around the first 3 weeks after diagnosis; interim measurement (T1) 6 weeks after baseline; post assessment measurement (T2) 12 weeks after baseline; follow-up measurement (T3) 6 month after baseline
  Physical activity enjoyment will be assessed with Physical Activity Enjoyment Scale - short version (PACES-S) to examine enjoyment levels related to physical activity.
  The questionnaire contains 4 questions. The score reaches from 0-16. The higher the score the greater the physical activity enjoyment.
Functional Appreciation, assessed via FAS | Baseline measurement around the first 3 weeks after diagnosis; interim measurement (T1) 6 weeks after baseline; post assessment measurement (T2) 12 weeks after baseline; follow-up measurement (T3) 6 month after baseline
  Functional Appreciation will be evaluated through the Functionality Appreciation Scale (FAS), which measures appreciation for the body's functional abilities.
  The score reaches from 7-35. The higher the score the greater the functional appreciation.
Motor abilities, assessed via Moon Test | Baseline measurement around the first 3 weeks after diagnosis; interim measurement (T1) 6 weeks after baseline; post assessment measurement (T2) 12 weeks after baseline; follow-up measurement (T3) 6 month after baseline
  Motor abilities will be assessed with the Moon Test, which measures across several key areas:
  Strength, speed, coordination, and flexibility will be evaluated with the Moon Test, which provides a comprehensive assessment of various motor skills in paediatric cancer patients. The Moon Test includes the following items: inserting pins, static stand, reaction test, stand and reach, medicine ball shot, sit to stand and hand grip strength.
  There is no overall score provided for the Moon Test.
Postural Balance, assessed via Force Plate | Baseline measurement around the first 3 weeks after diagnosis; interim measurement (T1) 6 weeks after baseline; post assessment measurement (T2) 12 weeks after baseline; follow-up measurement (T3) 6 month after baseline
  As a part of the motor abilities the postural balance will be assessed using a force plate to analyse body stability and balance control in bipedal, tandem, monopedal and a semi-tandem stand.
  The measurement variables are path length (cm) and the ellipse area (cm2). The higher the values the worse is the postural balance.
Physical Activity, assessed via BSA | Baseline measurement around the first 3 weeks after diagnosis; interim measurement (T1) 6 weeks after baseline; post assessment measurement (T2) 12 weeks after baseline; follow-up measurement (T3) 6 month after baseline
  Physical activity will be evaluated through the BSA (Measurement of physical and sports activity) to understand participants' activity levels. The BSA is a self-report questionnaire that assesses the frequency, intensity, and duration of physical and sports activities over a period of one month. Participants are asked to report their engagement in various activities, focused on structured sports, allowing for a comprehensive evaluation of their activity profile.
  The score ranges from 0 to 15 hours per week, with higher values indicating greater levels of physical activity. This measure captures both the intensity and time commitment to physical activities, providing insights into the participants' physical activity patterns.
Physical Activity, assessed via GSLTPAQ | Baseline measurement around the first 3 weeks after diagnosis; interim measurement (T1) 6 weeks after baseline; post assessment measurement (T2) 12 weeks after baseline; follow-up measurement (T3) 6 month after baseline
  Physical activity will be evaluated using the GSLTPAQ (Godin-Shephard Leisure-Time Physical Activity Questionnaire) to assess participants' typical activity levels during their leisure time. This questionnaire asks participants to report the frequency of mild, moderate, and vigorous physical activities they engage in over a typical week. Each category is weighted by its intensity to calculate a total Leisure Score Index (LSI), which provides an overall measure of physical activity.
  The theoretical score range for the Leisure Score Index (LSI) in the GSLTPAQ starts at 0 and typically extends up to 100, as most participants report values within this range. However, the scale is open-ended, allowing for higher scores depending on the frequency and intensity of reported physical activities. Higher scores indicate greater physical activity in leisure time.
Physical activity assessed via movement accelerometers | Only at interim measurement (T1) 6 weeks after baseline measurement for 7 consecutive days
  At T1(6 Weeks after baseline measurement) accelerometers and e-diaries will be used to quantify physical activity (PA) levels objectively (over a period of seven days) and to investigate children's affective experiences after sedentary behaviour and PA with a Ecological Momentary Assessment (EMA).
  Therefore, the Movisens Move4 accelerometers and study smartphones will be used.
  The Move 4 accelerometer, is a small three-axis sensor (movisens GmbH, Karlsruhe, Germany), which will be attached to the right hip, that captures body position and movement acceleration intensity.
Affective experiences, assessed via the Self-Assessment Manikin (SAM) | Only at interim measurement (T1) 6 weeks after baseline measurement for 7 consecutive days
  At T1(6 Weeks after baseline measurement) accelerometers and e-diaries will be used to quantify physical activity (PA) levels objectively (over a period of seven days) and to investigate children's affective experiences after sedentary behaviour and PA with a Ecological Momentary Assessment (EMA). Therefore, the Movisens Move4 accelerometers and study smartphones will be used.
  For the e-diaries the investigators will hand out smartphones and instruct the children to take them with them throughout seven days. Participants will be prompted to fill in the e-diary between 8am and 8pm, using a mixed sampling strategy.
  The Self-Assessment Manikin (SAM) will be used to measure the affective experience over the 7 days throughout the day on a Visual Analogue Scale (VAS).
Affective experiences and cancer related side effects, assessed via Present Functioning Visual Analogue Scales (PEDSQL VAS) | Only at interim measurement (T1) 6 weeks after baseline measurement for 7 consecutive days
  At T1(6 Weeks after baseline measurement) accelerometers and e-diaries will be used to quantify physical activity (PA) levels objectively (over a period of seven days) and to investigate children's affective experiences after sedentary behaviour and PA with a Ecological Momentary Assessment (EMA).
  Therefore, the Movisens Move4 accelerometers and study smartphones will be used.
  For the e-diaries the investigators will hand out smartphones and instruct the children to take them with them throughout seven days. Participants will be prompted to fill in the e-diary between 8am and 8pm, using a mixed sampling strategy.
  The Present Functioning Visual Analogue Scales (PEDSQL VAS) will be used to measure the affective experience and cancer related side effects over the 7 days throughout the day.
Current activity, assessed via e-diaries | Only at interim measurement (T1) 6 weeks after baseline measurement for 7 consecutive days
  At T1(6 Weeks after baseline measurement) accelerometers and e-diaries will be used to quantify physical activity (PA) levels objectively (over a period of seven days) and to investigate children's affective experiences after sedentary behaviour and PA with a Ecological Momentary Assessment (EMA).
  Therefore, the Movisens Move4 accelerometers and study smartphones will be used.
  For the e-diaries the investigators will hand out smartphones and instruct the children to take them with them throughout seven days. Participants will be prompted to fill in the e-diary between 8am and 8pm, using a mixed sampling strategy to get information about the current activity.
Muscle Mass (Body composition), assessed via Bioelectrical Impedance Analysis | Baseline measurement around the first 3 weeks after diagnosis; interim measurement (T1) 6 weeks after baseline; post assessment measurement (T2) 12 weeks after baseline; follow-up measurement (T3) 6 month after baseline
  Body composition will be assessed to understand the physical changes of the body. This includes the muscle mass measured by using a Bioelectrical impedance analysis.
Fat-Free Mass (Body composition), assessed via Bioelectrical Impedance Analysis | Baseline measurement around the first 3 weeks after diagnosis; interim measurement (T1) 6 weeks after baseline; post assessment measurement (T2) 12 weeks after baseline; follow-up measurement (T3) 6 month after baseline
  Body composition will be assessed to understand the physical changes of the body. This includes the fat-free mass measured by using a Bioelectrical impedance analysis.
Fat Mass (Body composition), assessed via Bioelectrical Impedance Analysis | Baseline measurement around the first 3 weeks after diagnosis; interim measurement (T1) 6 weeks after baseline; post assessment measurement (T2) 12 weeks after baseline; follow-up measurement (T3) 6 month after baseline
  Body composition will be assessed to understand the physical changes of the body. This includes the fat mass measured by using a Bioelectrical impedance analysis.
Feasibility of intervention, assessed via a self-developed questionnaire and semi-structured interviews | Baseline measurement around the first 3 weeks after diagnosis; interim measurement (T1) 6 weeks after baseline; post assessment measurement (T2) 12 weeks after baseline; follow-up measurement (T3) 6 month after baseline
  Feasibility of the intervention will be assessed to ensure it is practical, safe, and well-received by participants. This includes:
  A self-developed questionnaire and semi-structured interviews to evaluate whether the cognitively challenging physical activity intervention is feasible and motivating for the target group. The aim is to understand how manageable and engaging participants find the program.
Exercise adherence, assessed via exercise diary | During the intervention, expected to be on average 5 minutes
  Feasibility of the intervention will be assessed to ensure it is practical, safe, and well-received by participants. This includes exercise adherence. Exercise adherence will be tracked through an exercise diary to monitor participants' commitment to the program.
Feasibility of intervention | During the intervention, up to 6 months
  Feasibility of the intervention will be assessed to ensure it is practical, safe, and well-received by participants. This includes adverse events. Adverse events will be tracked within the exercise diary to monitor any physical or medical problems during intervention program.

OTHER OUTCOMES:
Demographic and clinical characteristics - Age | Baseline measurement around the first 3 weeks after diagnosis
  The investigators will collect data on demographic and clinical characteristics to understand the background of each participant. This includes the age of the participant.
  This information is needed for the overall information about the participant.
Demographic and clinical characteristics - Sex | Baseline measurement around the first 3 weeks after diagnosis
  The investigators will collect data on demographic and clinical characteristics to understand the background of each participant. This includes the sex of the participant.
  This information is needed for the overall information about the participant.
Demographic and clinical characteristics - Diagnosis | Baseline measurement around the first 3 weeks after diagnosis
  The investigators will collect data on demographic and clinical characteristics to understand the background of each participant. This includes the diagnosis o the participant.
  This information is needed for the overall information about the participant.
Demographic and clinical characteristics - Medical Treatment | Through individual study completion, an average of 6 to 8 months.
  The investigators will collect data on demographic and clinical characteristics to understand the background of each participant. This includes the medical treatment.
  This information is needed for the overall information about the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Valentin Benzing, Dr., Study Chair — University Bern; Eva Brack, Principal Investigator — University Children's Hospital Bern
Locations (1):
- Inselspital, Universitätsspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the published scientific articles will be made openly accessible on (BORIS, osf.io or Zenodo) after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The IPD will be available beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal will be able to assess the data. The data will be shared to achieve the aims of the provided proposal. BORIS, osf.io or Zenodo will be used to share the data after deidentification (text, tables, figures, and appendices).

REFERENCES:
- [Derived] Schneider AC, Hillebrecht L, Rehbein L, Schmid J, Pallivathukal S, von der Weid N, Furtwangler R, Brekenfeld RE, Greiner J, Schindera C, Brack EK, Benzing V. Smart exercise in pediatric oncology: enhancing executive functions through cognitively challenging physical activity- a non-randomized controlled trial. BMC Cancer. 2025 Dec 5;26(1):75. doi: 10.1186/s12885-025-15303-5. PMID 41351152
- See also: Exercise Recommendations for pediatric cancer patients — https://www.activeoncokids.org/betroffene/trainingsbroschuere-des-naok/